CLINICAL TRIAL: NCT01103115
Title: Can Calcium and Vitamin D Supplementation Improve Bone Mineral Density and Curve Progression in Girls With Adolescent Idiopathic Scoliosis?
Brief Title: Calcium + Vitamin D Supplementation for Low Bone Mass in Adolescent Idiopathic Scoliosis (AIS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHENG Chun-yiu Jack, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIS_Ca_VitD_01
Record Dates: First submitted 2010-04-05; First posted 2010-04-14 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; AIS; low bone mass; osteopenia; bone health; bone density
MeSH Terms: conditions — Scoliosis; Bone Diseases, Metabolic | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects in this group will take the placebo tablets
  Interventions: Dietary Supplement: Placebo
- Ca600mg+VitD400IU (Active Comparator): subjects receive a daily dose of 600 mg elemental calcium and 400 IU vitamin D3
  Interventions: Dietary Supplement: Calcium 600mg plus Vit D 400 IU
- Ca600mg+VitD800IU (Active Comparator): subjects receive a daily dose of 600 mg elemental calcium and 800 IU vitamin D3
  Interventions: Dietary Supplement: Calcium 600mg plus Vit D 800 IU

INTERVENTIONS:
Dietary Supplement: Calcium 600mg plus Vit D 400 IU — Daily supplementation with 600mg Calcium plus 400IU Vitamin D3
  Arms: Ca600mg+VitD400IU
Dietary Supplement: Calcium 600mg plus Vit D 800 IU — Daily supplementation with 600mg Calcium plus 800IU Vitamin D3
  Arms: Ca600mg+VitD800IU
Dietary Supplement: Placebo — placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Calcium and Vit D supplementation is effective for improving low bone mass in Girls with Adolescent Idiopathic Scoliosis (AIS).

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a prevalent condition mainly affecting females with disease onset at early puberty. It can lead to serious health problems and is associated with low bone mass which can persist with growth. Osteopenia is found to be an important prognostic factor for curve progression in AIS. Nutritional studies indicated AIS subjects had low dietary calcium intake. Evidences suggested that Vit D insufficiency could be present in AIS. Calcium and vitamin D supplementation can therefore be a viable treatment option for low bone mass in AIS subjects. The primary objective of this prospective randomized double-blinded placebo-controlled trial is to find out whether calcium and vitamin D supplementation can improve bone mineral density (BMD) in osteopenic AIS subjects. The secondary objective of this study is to evaluate whether the supplementation is effective in controlling curve progression in AIS.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 11-14 (Tanner stage < IV)
* Low BMD (z-score < 0 from age-matched population mean)
* Cobb's Angle greater or equal to 15°
* Presentation at the Scoliosis Clinic without prior treatment for low bone mass.

Exclusion Criteria:

* Scoliosis with any known etiology such as congenital scoliosis, neuromuscular scoliosis, scoliosis of metabolic etiology, scoliosis with skeletal dysplasia, or
* Patient with known endocrine and connective tissue abnormalities, or
* Patient with eating disorders or GI malabsorption disorders or
* Prior treatment for low bone mass before being recruited into the study.
* Patient currently taking medication that affects bone metabolism eg corticosterone or estrogen.

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 2-year time point
  To determine the effects of calcium and vitamin D intervention on improving bone mineral density of skeletally immature AIS girls with low bone mass.

SECONDARY OUTCOMES:
Curve severity | 2-year time point
  To determine the effects of calcium and vitamin D intervention on preventing curve progression of skeletally immature AIS girls with low bone mass.

CONTACTS AND LOCATIONS:
Overall Officials: Tsz-ping Lam, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- See also: Department of Orthopaedics and Traumatology, The Chinese University of Hong Kong — http://www.ort.cuhk.edu.hk/